CLINICAL TRIAL: NCT01991691
Title: Pilot Study for Tablet-based Questionnaire of Patient-reported Outcomes From Patients Undergoing Chemotherapy (TabPRO I)
Brief Title: Tablet-based Patient Reported Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Michael Mallmann, MD, Coordinating Investigator, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TabPRO I
Record Dates: First submitted 2013-11-17; First posted 2013-11-25 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Antineoplastic Agents
Keywords: Antineoplastic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tablet-based reported outcome (Experimental): With the start of chemotherapy until the end of the last cycle of chemotherapy the study participants have to document all signs of discomfort or changes to their overall coenesthesia in the tablet-based questionnaire.
  Interventions: Device: Tablet-based questionnaire

INTERVENTIONS:
Device: Tablet-based questionnaire — tablet-based patient reported outcomes (TabPRO)

SUMMARY:
This study is a single arm feasibility study. Patients that have been diagnosed with carcinoma and are undergoing chemotherapy have to document chemotherapy associated side effects on a regular basis by means of a tablet-based online questionnaire. Goal of the study is to find out if patients that are undergoing chemotherapy are willing to document chemotherapy associated side effects by means of a tablet-based online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients have to be ≥ 18 years of age
* written consent form and agreement to participate in the study
* patients that are able to follow the study instructions and that most likely will keep the required study appointments
* patients that have a histological confirmed carcinoma and are scheduled to undergo adjuvant or neoadjuvant chemotherapy of 6 to 8 cycles
* questions about chemotherapy associated side effects are composed in german. Therefore the study participants must have sufficient knowledge of the german language
* ECOG maximal level 2

Exclusion Criteria:

* patients that are younger than 18 years
* patients that don't agree to take part of the study
* patients that are not able to understand the scope, the meaning and the consequences of that clinical study
* patients that have a known or constant addiction to drugs or alcohol
* patients that suffer from blindness or dyslexia

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of Tablet-based questionnaire of PRO | 6 months
  Feasibility of Tablet-based questionnaire of PRO (>60% of patients answer >60% of questionnaires in the time frame of study duration)

SECONDARY OUTCOMES:
Answered questionnaires per patient | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mallmann, MD, Principal Investigator — Department of Obstetrics & Gynecology, University Hospital Bonn
Locations (3):
- Germany (3):
  - Department of Obstetrics & Gynecology, Evangelisches Krankenhaus Bergisch-Gladbach, Bergisch Gladbach
  - Department of Obstetrics & Gynecology, University Hospital Bonn, Bonn
  - Department of Obstetrics & Gynecology, University Hospital Cologne, Cologne

REFERENCES:
- [Background] Lipscomb J, Gotay CC, Snyder CF. Patient-reported outcomes in cancer: a review of recent research and policy initiatives. CA Cancer J Clin. 2007 Sep-Oct;57(5):278-300. doi: 10.3322/CA.57.5.278. PMID 17855485
- [Background] Dancey J, Zee B, Osoba D, Whitehead M, Lu F, Kaizer L, Latreille J, Pater JL. Quality of life scores: an independent prognostic variable in a general population of cancer patients receiving chemotherapy. The National Cancer Institute of Canada Clinical Trials Group. Qual Life Res. 1997 Mar;6(2):151-8. doi: 10.1023/a:1026442201191. PMID 9161115
- [Background] Garcia SF, Cella D, Clauser SB, Flynn KE, Lad T, Lai JS, Reeve BB, Smith AW, Stone AA, Weinfurt K. Standardizing patient-reported outcomes assessment in cancer clinical trials: a patient-reported outcomes measurement information system initiative. J Clin Oncol. 2007 Nov 10;25(32):5106-12. doi: 10.1200/JCO.2007.12.2341. PMID 17991929
- [Background] Basch E, Iasonos A, Barz A, Culkin A, Kris MG, Artz D, Fearn P, Speakman J, Farquhar R, Scher HI, McCabe M, Schrag D. Long-term toxicity monitoring via electronic patient-reported outcomes in patients receiving chemotherapy. J Clin Oncol. 2007 Dec 1;25(34):5374-80. doi: 10.1200/JCO.2007.11.2243. PMID 18048818
- [Background] Taenzer P, Bultz BD, Carlson LE, Speca M, DeGagne T, Olson K, Doll R, Rosberger Z. Impact of computerized quality of life screening on physician behaviour and patient satisfaction in lung cancer outpatients. Psychooncology. 2000 May-Jun;9(3):203-13. doi: 10.1002/1099-1611(200005/06)9:33.0.co;2-y. PMID 10871716
- [Background] Roizen MF, Coalson D, Hayward RS, Schmittner J, Thisted RA, Apfelbaum JL, Stocking CB, Cassel CK, Pompei P, Ford DE, et al. Can patients use an automated questionnaire to define their current health status? Med Care. 1992 May;30(5 Suppl):MS74-84. doi: 10.1097/00005650-199205001-00007. PMID 1583942